CLINICAL TRIAL: NCT04022369
Title: The Effects of an Exercise Empowerment Programme for Older Patients With Heart Failure: A Randomized Controlled Trial
Brief Title: The Effects of an Exercise Programme for Older Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Karaman (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Emine Karaman, Research Assistant Ms., PhD, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 12-9/7
Record Dates: First submitted 2019-07-08; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Old Age; Debility
Keywords: Aging; Randomized Controlled Trials (RCT); Nursing; Physical Activity
MeSH Terms: conditions — Heart Failure; Frailty; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The intervention group received 45-60 minute of individual training and a handbook for the exercise program was given. These patients were followed for a total of 12 weeks. The exercise program was developed by reviewing the literature part on physical activity for senior citizens with heart failure. Education program based on Empowerment model. Weekly motivational telephone interviews were conducted with the patients, and the home visits and telephone interviews were repeated when belived necessary. The purpose of the study were explained to all individuals involved in the study. Body movements, balance levels, exercise durations, and strengths of individuals before exercise program and after exercise program were evaluated. A booklet demonstrating the exercises was given to the patients to enhance their understanding, and they were allowed to ask questions about the exercise program during the training.
  Interventions: Behavioral: Exercise Group
- Control Group (No Intervention): The patients in the control group continued their standard treatment and care. Data collection forms were applied to the patients in the control group at the first month and 12 weeks after discharge. After the study was completed, all patients in the control group were provided with home-based exercise training booklets.

INTERVENTIONS:
Behavioral: Exercise Group — The intervention group received 45-60 minute of individual training and a handbook for the exercise program was given. These patients were followed for a total of 12 weeks. The weekly motivational phone calls structured according to the empowerment model and home visits when necessary were repeated. The exercise program was developed by reviewing the literature part on physical activity for senior citizens with heart failure. The program was established on evidence-based recommendations for the cardiac rehabilitation of patients with HF. Each session included warm-up and cool-down exercises, moderate walking, and balance exercises.
  Other Names: Control Group
  Arms: Exercise Group

SUMMARY:
Patients with heart failure have decreased exercise tolerance, balance problems, and fall risks. The purpose of this research was to investigate the effect of an exercise program based on the Empowerment Model for participants with heart failure. This randomized, controlled study including pre-test/post-test and the measurements were performed between January-November 2014 at a university hospital in Izmir, Turkey. Intervention group (n = 11) and control group (n = 10) participated in the research. The intervention group received 45-60 minute individual training and 12 weeks of individual follow-up. The weekly motivational phone calls structured according to the empowerment model and home visits when necessary were repeated. Patients in the control group did not receive any intervention except for their routine treatment. Data were collected before the education of exercise and after 12 weeks; sociodemographic data questionnaire, pedometer, accelerometer, Berg Balance Scale, HF Empowerment Scale, estimated weekly exercise monitoring form and exercise booklet had been utilised. The SPSS statistical package program was used to analyze the data.

DETAILED DESCRIPTION:
Patients with heart failure have decreased exercise tolerance, balance problems, and fall risks. The purpose of this research was to investigate the effect of an exercise program based on the Empowerment Model for participants with heart failure.

This randomized, controlled study including pre-test/post-test and the measurements were performed between January-November 2014 at a university hospital in Izmir, Turkey. Intervention group (n = 11) and control group (n = 10) participated in the research. The intervention group received 45-60 minute individual training and 12 weeks of individual follow-up. The weekly motivational phone calls structured according to the empowerment model and home visits when necessary were repeated. Patients in the control group did not receive any intervention except for their routine treatment. Data were collected before the education of exercise and after 12 weeks; sociodemographic data questionnaire, pedometer, accelerometer, Berg Balance Scale, HF Empowerment Scale, estimated weekly exercise monitoring form and exercise booklet had been utilised. The SPSS statistical package program was used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* were aged 60 years or older
* independent
* literate
* able to communicate verbally
* participating voluntarly in the study

Exclusion Criteria:

* were having a diagnosis of psychiatric illness
* a visual or auditory impairment
* previously participated in another exercise program
* any contraindication to exercise (uncontrolled arrhythmia, hypertension and metabolic illness, ejection fraction)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2015-07-06 (Actual)

PRIMARY OUTCOMES:
Group (empowerment evaluation scale assessment) | 3 months
  Old patients were observed and evaluated daily activities during 12 weeks. The exercise program was established on evidence-based recommendations for patients with Heart Failure (HF). Empowerment level of individuals before and after exercise program were evaluated. Empowerment is a model aiming to protect patients' rights and develop the quality of care. This model is aimed at giving individuals a feeling of success and improving their self image, and is intended to make necessary lifestyle changes easier and more lasting. Subscales of the empowerment are "Managing the Psychosocial Aspects of Heart Failure", "Assessing Dissatisfaction and Readiness to Change" and "Setting and Achieving Heart Failure Goals". The Scale evaluated has 28 items and five-way likert-type. Scores range from 28 to 140, scores of 28-65 classified as low, 66-103 as medium, and 104-140 as high.

SECONDARY OUTCOMES:
Control Group (empowerment evaluation scale assessment) | 3 months
  The patients in the control group continued their routine treatment and daily living activities. These patients were observed and evaluated daily activities during 12 weeks. Empowerment level of the individuals before and after 12 weeks were evaluated. Empowerment is a model aiming to protect patients' rights and develop the quality of care. This model is aimed at giving individuals a feeling of success and improving their self image, and is intended to make necessary lifestyle changes easier and more lasting. Subscales of the empowerment are "Managing the Psychosocial Aspects of Heart Failure", "Assessing Dissatisfaction and Readiness to Change" and "Setting and Achieving Heart Failure Goals". The Scale evaluated has 28 items and five-way likert-type. Scores range from 28 to 140, scores of 28-65 classified as low, 66-103 as medium, and 104-140 as high.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Çiçek FADILOĞLU, Emertus, Study Director — Ege University

IPD SHARING:
Plan to Share IPD: Yes
The intervention group received 45-60 minute of individual training and a handbook for the exercise program was given. These patients were followed for a total of 12 weeks. The exercise program was developed by reviewing the literature part on physical activity for senior citizens with heart failure. Education program based on Empowerment model. Weekly motivational telephone interviews were conducted with the patients, and the home visits and telephone interviews were repeated when belived necessary. The purpose of the study were explained to all individuals involved in the study. Body movements, balance levels, exercise durations, and strengths of individuals before exercise program and after exercise program were evaluated. A booklet demonstrating the exercises was given to the patients to enhance their understanding, and they were allowed to ask questions about the exercise program during the training.
Time Frame: 3 months
Access Criteria: The purpose of this research was to investigate the effect of an exercise program based on the Empowerment Model for participants with heart failure.